CLINICAL TRIAL: NCT05444140
Title: A Theory-guided Health Coaching Programme for Middle-aged Adults With Cardiometabolic Risk to Improve Health Promoting Behaviours: a Feasibility Study
Brief Title: A Feasibility Study of a Health Coaching Programme for Middle-aged Adults With Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zoe Ching Man Kwok, Lecturer, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Health coaching midlife pilot
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cardiometabolic Disease; Health Coaching; Middle-aged Adults; Primary Prevention
Keywords: cardiometabolic disease; feasibility study; health coaching; middle-aged adults; primary prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Health coaching
  Interventions: Behavioral: Health coaching

INTERVENTIONS:
Behavioral: Health coaching — The health coaching programme includes four monthly health coaching sessions for three months.

SUMMARY:
Cardiometabolic disease has been an increasing trend globally and remains the major cause of morbidity and mortality. Health coaching, a process of goal-oriented and client-centered partnership that is health-focus and through client enlightenment and empowerment, are generally effective for chronic disease management and prevention of complication. However, there is inconclusive result on the effects of health coaching in the primary prevention of cardiometabolic diseases. Therefore, this study aimed to assess the feasibility and acceptability of a theory-guided health coaching programme for middle-aged adults with cardiometabolic risk.

DETAILED DESCRIPTION:
A single group pretest-posttest feasibility study was conducted. The health coaching programme included four monthly health coaching sessions for three months. Feasibility of the study was measured by eligibility rate, enrollment rate, adherence rate, and attrition rate. Intervention acceptability was measured by satisfactory survey after completion of health coaching intervention. Feasibility of outcome measures was measured by the completion of outcome measures assessment at baseline and 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-64 years;
* have a non-laboratory INTERHEART risk score (IHRS) of 16 or higher;
* can communicate in Cantonese;
* able to give informed consent.

Exclusion Criteria:

* previous diagnosis of transient ischemic attack, stroke, myocardial infarction, atrial fibrillation, coronary heart disease, heart failure, dementia, chronic renal failure and diabetes;
* currently on medication to control hyperlipidemia, diabetes or hypertension;
* with eye or retinal disease;
* diagnosis of terminal disease with an expected life expectancy less than 12 months;
* currently participating in any other clinical trial;
* currently participating in any other structured lifestyle-based or exercise-based programme.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of study | at baseline
  eligibility rate, enrolment rate
Feasibility of study | at 3 months after enrolment
  adherence rate
Feasibility of study | at 3 months after enrolment
  attrition rate
Feasibility of study | at 6 months after enrolment
  attrition rate
Intervention Acceptability | at 3 months after enrolment
  Participants' satisfaction survey
Feasibility of outcome measures assessment | at baseline
  completion rate of a battery of outcome measures assessment (including (1) health promoting behaviours measures using Health Promoting Lifestyle Profile II (HPLP II); (2) cardiometabolic risk measured using non-laboratory INTERHEART risk score and the Automatic Retinal Image Analysis (ARIA)-stroke model; (3) self-efficacy of adopting health-promoting behaviours measured using Diabetes Mellitus Type II Self Efficacy Scale; (4) psychological distress measured using the Chinese version of the shorter version of Depression Anxiety Stress Scales (DASS); (5) sleep quality measured using the Chinese version of the Pittsburg Sleep Quality Index; (6) physical activity level measured using the International Physical Activity Questionnaire-Chinese (IPAQ-C); and (7) physiological parameters, including blood pressure, body mass index (BMI), waist-hip-ratio (WHR) and point of care blood test for glucose, lipid and urate level)
Feasibility of outcome measures assessment | at 6 months after enrolment
  completion rate of a battery of outcome measures assessment (including (1) health promoting behaviours measures using Health Promoting Lifestyle Profile II (HPLP II); (2) cardiometabolic risk measured using non-laboratory INTERHEART risk score and the Automatic Retinal Image Analysis (ARIA)-stroke model; (3) self-efficacy of adopting health-promoting behaviours measured using Diabetes Mellitus Type II Self Efficacy Scale; (4) psychological distress measured using the Chinese version of the shorter version of Depression Anxiety Stress Scales (DASS); (5) sleep quality measured using the Chinese version of the Pittsburg Sleep Quality Index; (6) physical activity level measured using the International Physical Activity Questionnaire-Chinese (IPAQ-C); and (7) physiological parameters, including blood pressure, body mass index (BMI), waist-hip-ratio (WHR) and point of care blood test for glucose, lipid and urate level)

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Kwok, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwok ZC, Tam HL, Zee BC, Lo SW, Tang FW, Tao A, Chan HY. A protection motivation theory-guided telehealth coaching program for middle-aged adults with cardiometabolic risk: A feasibility trial. BMC Public Health. 2025 Mar 24;25(1):1120. doi: 10.1186/s12889-025-22238-w. PMID 40128717